CLINICAL TRIAL: NCT06618833
Title: Medical and Sociological Characterization of the Population of Patients Admitted for a First Ablation of Atrial Fibrillation in the Occitanie Ouest Region
Acronym: CAMS-AFA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/23/0539; 2023-A02755-40 (Registry Identifier: ID-RCB Number)
Record Dates: First submitted 2024-09-23; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Fibrillation, Atrial
Keywords: Medical and Sociological Characterization of the Population; Global Promis Questionnaire
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient admitted for first atrial fibrillation ablation (Experimental)
  Interventions: Other: Collection of medical data; Behavioral: Collection of global health elements; Behavioral: PROMIS global questionnaire; Behavioral: Collection of sociological data

INTERVENTIONS:
Other: Collection of medical data — Collection of medical data focused on the history of atrial fibrillation by the principal investigator
Behavioral: Collection of global health elements — Collection of global health elements (physical and mental) by the principal investigator by discussion with the patient
Behavioral: PROMIS global questionnaire — The patient completes the global PROMIS questionnaire which collects data on their overall health.
  The questionnaire consists of 10 questions about the patient's overall health, and for each question, the patient has a possible choice of 5 answers varying between different propositions depending on the question:
  Excellent to poor or Totally to not at all, or Always to never or None to very intense
Behavioral: Collection of sociological data — Collection of patient sociological data (territorial, economic, professional, ethnic) by the principal investigator

SUMMARY:
Atrial fibrillation is the most common arrhythmia with a prevalence of 1 to 4% and constitutes a major health problem both on an individual level (impaired quality of life, heart failure, stroke, hospitalization, excess mortality) and collective level (cost, use of resources).

Non-medical determinants influence health, particularly its cardiovascular component, but have been little studied in the context of Atrial fibrillation. The rare studies addressing the subject suggest that they impact the incidence of the disease and the occurrence of its complications. Certain social and sociological characteristics are also associated with less access to the various recognized therapies, whether medicinal or invasive. This is the case for Atrial fibrillation ablation, which has nevertheless demonstrated its usefulness in reducing the Atrial fibrillation burden, in reducing symptoms and hospitalizations and for certain populations (heart failure) a decrease in mortality.

Essien et al in a literature review report that non-Caucasian and low-income people have less access to Atrial fibrillation ablation. Non-Caucasian populations are also under-represented in interventional clinical studies on Atrial fibrillation. If the level of education (health literacy), geographic origin (rural vs. urban) and the level of isolation affect the occurrence of Atrial fibrillation and its natural history, including complications, the authors do not mention any specific study that has evaluated their role in access to ablation.

A Norwegian national analysis (Olsen) based on data from the health system, therefore exhaustive, evaluated the characteristics of patients suffering from Atrial fibrillation and having benefited from ablation compared to the characteristics of patients treated medically. Patients with the highest levels of education and income are the most likely to be treated by ablation. Women, especially at younger ages, have less access to ablation. The authors also found significant differences between the different territorial subdivisions of the country.

DETAILED DESCRIPTION:
There are therefore arguments highlighting the role of non-medical determinants in the management of Atrial fibrillation by ablation. However, they come from studies from countries (USA, Canada, Norway) whose characteristics may not be universally applicable. The investigator can also question the lack of detail of the data that come from national databases and which lack variables to precisely characterize this population. The investigator therefore wish to carry out an observational study aimed at defining on a medical, sociological, economic and territorial level the population having access to Atrial fibrillation ablation in the Occitanie Ouest population basin (represented by the former Midi-Pyrénées region). The data will come from the only two centers performing this type of intervention, the Pasteur clinic and the Toulouse University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted for first ablation of Atrial Fibrillation

Exclusion Criteria:

* Patients under 18 years of age
* Pregnancy
* No coverage by the French health system
* Refusal to consent
* History of left atrium ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Collection of medical and sociological data from the population of patients admitted for a first Atrial Fibrillation Ablation | 2 months
  Collection of medical data (cardiological, comorbidities, physical and mental health via PROMIS global questionnaire) and sociological data (territorial, economic, professional, ethnic, family). The PROMIS GLOBAL questionnaire is a questionnaire to collect data on the patient's general health. It is presented in 10 questions. The answers can vary between "Excellent to Poor", "Totally to Not at All", "Never to Always" or even "None to Very Intense"

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre DUPARC, MD, Principal Investigator — University Hospital, Toulouse
Locations (2):
- France (2):
  - Clinique Pasteur, Toulouse
  - Rangueil Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: No